CLINICAL TRIAL: NCT02860832
Title: The Relationships of Cyber-bullying and Bullying With Self-esteem, Depression and Suicidal Ideation Among Taiwanese Adolescents: Mixed Method Study
Brief Title: The Relationships of Cyber-bullying and Bullying With Mental Health Among Taiwanese Adolescents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201601074RIND
Record Dates: First submitted 2016-06-23; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Depression
Keywords: Cyberbullying; Traditional bullying; Depression
MeSH Terms: conditions — Depression; Cyberbullying

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Background and significance: Though the problem of bullying among adolescents is evidently increasing and of a serious social concern, it is often undetected until serious outcomes have surfaced. In recent years, along with the rapid expansion of the Internet, social network services (SNS) and smart phones, "cyber-bullying" has been growing. Compared to the traditional bullying, cyberbullying is unique in nature and potentially more hazardous in terms of invisibility, lack of control, where it enables communication with a broad range of people at any time and place.

To explore deeper understanding of the magnitude and the impact of the bullying among adolescents in Taiwan to inform public policy and future health intervention programs may be beneficial not only to Taiwan but also to Asia as a whole. Many Asian countries now suffer the similar problems of bullying among adolescents, since these countries share similar characteristics of development (spread of internet, SNSs and smart phones).

Goal and objectives: This study aims to explore Taiwanese adolescents' experiences, perceptions, opinions and mental health regarding cyberbullying and traditional bullying to inform the development of questionnaire in the quantitative phase of mixed methods study.

Study design: A qualitative study design with in depth interviews will be adopted.

Target population and study setting: Senior high school students will be recruited from Taipei city, Taiwan.

Sample size and sampling method: Participants will be sampled by convenience sampling until thematic saturation is attained, probably around 50 students.

Data collection: Face-to-face in-depth interview with semi-structured questionnaire will be used.

Data analysis: All interviews will be voice-recorded, transcribed, analyzed by thematic analysis procedure. Analysis process will include familiarization, coding, searching for themes, reviewing the themes, defining, naming themes and writing up or weaving the analytic narrative. Triangulation and supervision will also ensure credibility and balance in the process.

DETAILED DESCRIPTION:
Background and significance: Though the problem of bullying among adolescents is evidently increasing and of a serious social concern, it is often undetected, overlooked and noticeable only after serious outcomes have surfaced. In the recent years, along with the rapid expansion of internet, social network services (SNS) and smart phones, bullying through such electronic means, "cyber-bullying", has been growing. Compared to the traditional bullying cyberbullying is unique in nature and potentially more hazardous in terms of invisibility, lack of control, where it enables communication with a broad range of people at any time and at any place. This study is based on mixed methods study. The investigators hope that the investigators study could contribute to the deeper understanding of the magnitude and impact of the bullying among adolescents in Taiwan and to inform public policy and future health intervention programs which may be beneficial not only to the Taiwan but to Asia, as a whole, as many Asian countries now suffer the similar problems of bullying among adolescents as the countries share similar characteristics of development (spread of internet, SNSs and smart phones) having resembling lifestyle and values.

Study purpose: The purpose of this study is to investigate the prevalence of traditional bullying and cyberbullying and the association between cyber-bullying and traditional bullying with mental health among Taiwanese adolescents.

Study design: A mixed methods research design with qualitative study followed by quantitative study will be used in this research. Senior high school students will be included in Taiwan. For qualitative phase of this study, purposive sampling will be used to recruit students. For the quantitative phase of the study, sampling will be conducted by probability proportionate to size sampling procedure. For the qualitative phase of this study, in depth interview will be used to develop the quantitative questionnaire. An anonymous questionnaire developed from qualitative will be used to measure the variable of self-esteem, depression, suicidal ideation, traditional bullying and cyberbullying.

Data analysis: For qualitative study, all interviews will be voice-recorded, transcribed, analyzed by thematic analysis procedure. Quantitative data will be statistically analyzed by using SAS software. Descriptive data will be calculated for all variables. Multiple regressions will be performed to understand the relationship between socio-demographic variables, cyberbullying, traditional bullying, self-esteem, depression and suicidal ideation which separated by gender.

ELIGIBILITY:
Inclusion criteria

* The 16-18 aged high school students now studying in Taipei will be recruited in this study.

Exclusion criteria

* Students who are attending schools at night, since it's difficult to require them to participate in our research.
* Students who are studying in special educational schools for mentally handicapped because they will be unable to be interviewed and complete questionnaires. Also those who failed to obtain parental consents and individual consents will be excluded from the study.

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Senior high school students will be recruited from Taipei city, Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
The students of depression will be measured by questionnaire. | one year
The students of suicidal ideation will be measured by questionnaire. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Chuan Chan, Principal Investigator — Department of public health, college of public health, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No